CLINICAL TRIAL: NCT04631042
Title: An Observational Study of the Developing Brain, Impulsivity and Compulsivity
Brief Title: Developing Brain, Impulsivity and Compulsivity
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200147; 20-HG-0147
Record Dates: First submitted 2020-11-14; First posted 2020-11-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Typical Development; Obsessive Compulsive Disorder; Conduct Disorder; Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder
Keywords: Neurodevelopmental disorder; Twin; Natural History; Heritability; Glutamate; developmental trajectory; Brain Connectivity
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Conduct Disorder; Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- impulsive compulsive: Individuals between 6 and 80 years of age with a wide range of impulsivity/compulsivity behaviors - ranging from normal to mildly/extremely impaired.

SUMMARY:
Background:

Impulsivity is acting 'without thinking.' Compulsivity is being overly inflexible. People vary in how impulsive or compulsive they are. Extreme versions of these behaviors play a role in mental disorders. Researchers want to study changes in the brain to learn more about these behaviors. Differences in genes may also play a role.

Objective:

To learn about genetic & brain features that explain why levels of impulsivity and compulsivity vary across people.

Eligibility:

People ages 6 - 80

Design:

Participants will be screened with a medical history and medical record review.

Participants will talk about their mental and behavioral development. They may discuss topics like drug use and sexual activity. They will complete surveys about their compulsivity and impulsivity. Parents of child participants may also complete these surveys.

Participants may take memory, attention, and thinking tests. They may give blood or saliva samples for gene studies and they may give blood to make induced pluripotent stem cells. Participants may have their face and irises photographs taken.

Participants may have a magnetic resonance imaging scan. It will take pictures of their brain. The scanner is shaped like a cylinder. Participants will lie on a table that slides in and out of the scanner. A coil will be placed over their head. They will lie still, watch a movie, and play a game.

Participants may ask family members to join the study. Researchers are particularly interested in recruiting twin pairs to the study.

Participants under age 25 may repeat these tests every 1-2 years until they turn 25 or until the study ends. For those over age 25, participation will last less than 1 month.

DETAILED DESCRIPTION:
Study Description:

Many neuropsychiatric disorders have extreme impairing impulsivity and compulsivity behaviors at their core. We hypothesized that the development of symptoms of impulsivity and compulsivity during childhood/adolescence and early adulthood will be associated with atypical trajectories of brain features including cortical glutamate (the main excitatory neurotransmitter) and functional/structural brain connectivity. Additionally, we hypothesize that cortical glutamate will be under genetic control (i.e., heritable) and that common genetic variant risk for disorders characterized by extreme impulsivity (e.g., attention deficit hyperactivity disorder) and by extreme compulsivity (e.g., obsessive compulsive disorder, autism spectrum disorder) will also be associated with atypical cortical glutamate trajectories. To elucidate the relationships between the developing brain, compulsivity/impulsivity and genomics, we will collect clinical assessments including clinician-led interviews, neurobehavioral assessments, neuroimaging data, and genomic samples using 1) a prospective longitudinal design to answer developmental hypotheses; 2) a twin design to assess heritability hypotheses.

Objectives:

Primary Objective:

A) To assess the effects of impulsivity and compulsivity on the developmental trajectories of cortical glutamate.

B) To determine the heritability of cortical glutamate.

Secondary Objectives:

A) To establish the reliability of glutamate measurements.

B) To examine the impact of atypical glutamate levels on developing structural and functional connections within the fronto-striatal circuits.

C) To assess within twin pair differences in neurodevelopmental markers (cortical glutamate, structural/functional MRI) in relation to differences in symptom domains.

Endpoints:

Primary Endpoint:

A) Age-related change in cortical glutamate levels and its moderation by individual differences in levels of impulsivity and compulsivity.

B) Heritability of cortical glutamate (proportion of variance explained by additive genetic factors).

Secondary Endpoints:

A) 1) Glutamate levels estimated at 3 Tesla at short intervals to establish test-retest reliability.

2) Glutamate levels estimated at both 3 Tesla and 7 Tesla (cross scanner validation).

B) Measures of the brain's structural and functional connectivity.

C) Within twin-pair differences in neurodevelopmental markers symptom domains (impulsivity/compulsivity).

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Must be between 6 and 80 years of age.
3. Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Cognitively not capable of performing study procedures or lack of capacity to provide informed consent. Indications of a lack of cognitive capacity could include a known full-scale IQ under 70, or a history from the screening interview that implies global intellectual disabilities (e.g., placement in a school for children with intellectual disability etc.)
2. Very premature birth (i.e., birth before 32 weeks of gestational age).
3. Any known brain abnormalities (e.g., tumor, periventricular leukomalacia, microcephaly) or history of medical conditions known to affect cerebral anatomy (e.g., epilepsy, history of stroke, head injury with a loss of consciousness of one hour or more).
4. Psychotic disorders (including schizophrenia, psychosis not otherwise specified).
5. Dementia, or other conditions that, in the opinion of the investigators, would impede compliance or possibly hinder completion of the study.
6. Pregnant women.
7. Any other medical or psychiatric condition that in the opinion of the PI may confound study data/assessments.

Additional exclusion criteria for optional MRI procedure:

1. Individuals who are not able to receive an MRI (e.g., metal bioimplants, claustrophobia, inability to lie flat on their backs, pregnant women, and any other contraindications for MRI scanning according to the NMR Center MRI safety guidelines).

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals between 6 and 80 years of age with a wide range of impulsivity/compulsivity behaviors - ranging from normal to mildly/extremely impaired - will be recruited. No specific demographic groups will be targeted. Recruitment will be mainly done in the District of Columbia/Maryland/Virginia area, however some participants might travel from elsewhere.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Glutamate concentration measured using Magnetic Resonance Spectroscopy | Yearly if possible
  Age-related change in cortical glutamate levels and its moderation by individual differences in levels of impulsivity and compulsivity.
Heritability of cortical glutamate (proportion of variance explained by additive genetic factors). | Baseline
  Degree to which glutamate levels are under genetic control.

SECONDARY OUTCOMES:
Structural and functional connectivity | Yearly if possible
  Structural and functional connectivity measured throughout development using Magnetic Resonance Imaging.
Glutamate levels | weeks to months
  Glutamate measurement at 7 Tesla is now the gold standard for glutamate measurements, against which we will compare measurements at 3 Tesla.
Differences in glutamate levels and other neurodevelopmental markers within twin pairs. | Yearly if possible
  Differences in twin characteristics will be measured through clinical symptom assessment, biomarkers, Magnetic Resonance Imaging, neuropsychological testing, and questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya J White, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified medical information will be placed in a NIH repository (e.g., Biomedical Translational Research Information System (BTRIS)) in accordance to NIH policies. We will also share genomic and phenotypic data in controlled access databases such as dbGAP (database of Genotypes and Phenotypes). Other databases may be used as approved by NIH for the sharing of de-identified data.
Supporting Information: Study Protocol
Time Frame: The timeline for data sharing will follow the NHGRI Genomic Data Sharing Policy. Currently data is deposited following IRB review once the study data collection is complete and the data has undergone quality control steps.
Access Criteria: Access requests for specific research purposes using NIH controlled-access data are reviewed by NIH Data Access Committees (DACs).

REFERENCES:
- [Background] Ziegler G, Hauser TU, Moutoussis M, Bullmore ET, Goodyer IM, Fonagy P, Jones PB; NSPN Consortium; Lindenberger U, Dolan RJ. Compulsivity and impulsivity traits linked to attenuated developmental frontostriatal myelination trajectories. Nat Neurosci. 2019 Jun;22(6):992-999. doi: 10.1038/s41593-019-0394-3. Epub 2019 May 13. PMID 31086316
- [Background] Naaijen J, Lythgoe DJ, Amiri H, Buitelaar JK, Glennon JC. Fronto-striatal glutamatergic compounds in compulsive and impulsive syndromes: a review of magnetic resonance spectroscopy studies. Neurosci Biobehav Rev. 2015 May;52:74-88. doi: 10.1016/j.neubiorev.2015.02.009. Epub 2015 Feb 21. PMID 25712432
- [Background] Fineberg NA, Chamberlain SR, Goudriaan AE, Stein DJ, Vanderschuren LJ, Gillan CM, Shekar S, Gorwood PA, Voon V, Morein-Zamir S, Denys D, Sahakian BJ, Moeller FG, Robbins TW, Potenza MN. New developments in human neurocognition: clinical, genetic, and brain imaging correlates of impulsivity and compulsivity. CNS Spectr. 2014 Feb;19(1):69-89. doi: 10.1017/S1092852913000801. PMID 24512640
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-HG-0147.html